CLINICAL TRIAL: NCT06648967
Title: Hydrogen Breath Test Results After Consuming Fructose at Baseline and After Protein Supplementation
Brief Title: Impact of Different Carbohydrate Feedings on a Hydrogen Breath Curve and Self-reported Gastrointestinal Complaints
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Floris Wardenaar, Assistant Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00020453
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Quality of Life
Keywords: participants; healthy subjects; women; men; malabsorption syndrome
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Malabsorption Syndromes | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseline exercise tests with carbohydrate feeding and after supplementation (Experimental): This arms includes the assessment for difference between two different boluses of carbohydrate after a hiking test in the heat on fructose malabsorption measured by determining a hydrogen breath curve, as well as taking multiple self-reported gastrointestinal symptom ratings during exercise test 1 and 2. In addition, this arm will assess hydrogen breath response and gastrointestinal symptom ratings (using one of the previously determined carbohydrate boluses) after supplementing a multi-ingredient whey protein for 3 weeks, followed by 2 more weeks of supplementation.
  Interventions: Dietary Supplement: Supplementation with a multi-ingredient whey supplement

INTERVENTIONS:
Dietary Supplement: Supplementation with a multi-ingredient whey supplement — Malabsorption of two different fructose boluses at baseline and after 3 and 5 weeks of multi-ingredient whey supplementation.

SUMMARY:
GI distress is widely prevalent among athletes, ranging from 30 to 90% in recreationally and professionally active athletes. As the recipient of nutrients, the gastrointestinal (GI) tract plays an important role in athleticism. The following pilot project aims to better understand if a fructose load after hiking under heat stress will result in a meaningful hydrogen breath elevation as a marker for malabsorption in healthy participants, and if supplementation of a multi-ingredient fermented whey supplement will result in a different hydrogen breath response rate after a heat stress hiking test.

DETAILED DESCRIPTION:
The present study aims to examine the difference between two different boluses of carbohydrate after a hiking test in the heat on fructose malabsorption measured by determining a hydrogen breath curve, as well as taking multiple self-reported gastrointestinal symptom ratings.

In addition, the study aims to evaluate the difference in hydrogen breath response and gastrointestinal symptom ratings (using one of the previously determined carbohydrate boluses) after supplementing a multi-ingredient whey protein for 3 weeks, followed by 2 more weeks of supplementation.

The objective of the study is to answer following questions:

Question 1: Does treadmill hiking in the heat combined with a glucose-fructose feeding (i.e. ration 2:1 or 1:2) result in different hydrogen breath malabsorption curves and GI symptoms.

Question 2: Is there a difference in hydrogen breath test curves and self-reported gastrointestinal symptom ratings over time, after 3 and 5 weeks of supplementation, when consuming a multi-ingredient whey supplement compared to baseline.

No study procedures will start until informed consent has been obtained.

The familiarization: If participants meet all the inclusion criteria and choose to participate, participants will start with the familiarization to get a better feeling of the type of exercise they need to perform. Participants will perform an "Ebbeling Submax Test", a two-stage walking protocol lasting ~10 minutes. After this VO2max is determined from the steady state heartrate (HR) and speed following the last 4 minutes of the second stage at 5% grade. Steady state HR is defined as over 120 bpm and ±5 bpm range over at least 2 minutes.

Test protocol: The night prior to each exercise test date, the participant will be asked to consume a standardized, low-fiber meal which will be provided to them. After 10pm, participants will be asked not to consume any calorie containing items and to only consume water. Participants will also be asked to avoid exercising the day prior to testing. The day of the test, participants will arrive fasted, and they will perform a 60-minute hiking protocol in a warm environment. The exercise consists of hiking on a treadmill in a warm environment (>30-35°C), while reaching an exercise intensity of 70% ±5 bpm of the subject's HR max (calculated by the Karvonen method as described below). Which is an intensity in which the subject has an elevated breathing frequency but is still able to talk. The treadmill has a 5% incline, and participants will start at a speed informed by their Ebbeling test results, after this each minute the speed will be increased with 0.5 mph until the heartrate reflects the target HR range, in case walking speed is maxed out treadmill incline can be altered as well. Heart rate and speed will be continuously monitored, if speed needs to be adjusted at a later phase during the protocol (because heartrate is not within the targeted HR-range) this will be recorded to allow for exact copying the protocol during the next exercise sessions. The exercise will be divided in 3 blocks of 20 minutes during which the participants work towards reaching their 70% HR max during an 18-minute period, followed with 2 minutes active rest if needed before the next block. The carbohydrate feeding will consist of 3 carbohydrate gels with ~25 grams of carbohydrate with a 2:1 ratio glucose and fructose during, followed by 500 mL water during test 1, and consumption of 25 grams of glucose in 100 mL at the start of test 2 followed by 50 grams of fructose after the test mixed in 400 mL, no food will be provided after the heat stress test, but water can be consumed ad libitum. Heart rate will be monitored using a heart rate monitor attached via chest strap. Monitor will be placed by the participant beneath all clothing with the monitor at chest level (xyphoid process) with guidance from the research team. If the participant requests help, a research team member will assist.

Hydrogen Breath Analysis: Hydrogen measurements will be issued at baseline (-65min), post-exercise (0min), and with 30-min intervals post-exercise at 30/60/90/120/150 and 180 min. Hydrogen breath analysis is a minimally invasive procedure which requires the participant to breath normally but exhale into a gas sample bag until the 250mL bag is filled.

Gastrointestinal Distress: Accompanying the hydrogen breath test at -65min, 0min, 60min, 120min and 180mi, a GSRS questionnaire will also be given. The GSRS consists of 15 items and typically assesses GI complaints in the seven days before survey administration, however, instructions will be modified to request symptoms experienced at the time of administration. The GSRS will be administered digitally in this study and will require less than 5 minutes to complete. The 15 items (1: Upper abdominal pain; 2: Heartburn; 3: Acid reflux; 4: Hunger pains; 5: Nausea; 6: Rumbling in the stomach; 7: Bloated; 8: Burping; 9: Passing gas or flatus; 10: Constipation; 11: Diarrhea; 12: Loose stools; 13: Hard stools; 14: Urgent need to defecate; 15: Incomplete emptying of bowels) assessed the extent of discomforts of GI symptoms based on a 7-point Likert scale, where higher scores reflect more severe discomforts. A total score with no complaints would result in 15 points, whereas the maximal score would result in 105 points.

Baseline testing (exercise test 1 and test 2): Participants will be scheduled for 2 separate test visits including a 60 min hiking test, followed by 3 hours of hydrogen breath data and gastrointestinal symptoms data collection. The two visits set one week apart will be completed. No supplementation between these visits will be consumed and participants will be advised to mimic exercise and diet the day prior to testing. On both visits, participants will arrive fasted and will complete the testing protocol as described below. At the end of the second visit, instructions for the 3-week supplementation will be given to the participants and the product will be sent home with them.

Testing after supplementation (exercise test 3 and test 4): After these baseline visits, a 3-week protein supplementation protocol will be completed followed by again a test visit, followed by an additional 2-week protein supplementation protocol and a final test visit. The commercially available protein supplement (Biotis® Fermentis), is a multi-ingredient fermented whey supplement with 8 g of protein and 4 g of soluble fiber (galactooligosaccharides) per serving.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects living in the United States.
* Women/Men aged between 18-60 years (50-50%).
* BMI value between ≥18.5 and ≤ 30 kg/m2.
* No physical limitations (i.e., able to perform all activities associated with daily living in an independent manner).
* Written informed consent.
* Completed PAR-Q+ without any "yes" responses.
* If currently using chronically or intermittently, willing to stop taking pre- and probiotics beginning 1 month prior to and throughout data collection.
* If currently using chronically or intermittently, willing to stop using laxatives or fiber supplements, antacids and prokinetics beginning 1 month prior to and throughout data collection.

Exclusion Criteria:

* Smoking.
* Clinical or self-perceived lactose intolerance.
* Clinical or self-perceived milk protein allergy.
* Diagnosed GI tract disorders or diseases.
* Musculoskeletal disorders.
* Diagnosed metabolic disorders (such as diabetes).
* Use of any medications known to affect protein metabolism (i.e., corticosteroids, non-steroidal anti-inflammatories, or prescribed acne medications).
* Chronic use of gastric acid suppressing medication or anti-coagulants.
* Chronic use of anti-inflammatory medication.
* Unwilling to stop taking pre- and probiotics beginning 1 month prior to and throughout data collection.
* Unwilling to stop using laxatives or fiber supplements, antacids and prokinetics beginning 1 month prior to and throughout data collection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Hydrogen breath curve | Measurements will be taken at -65 min before exercise, directly after exercise at 0 min, and at 30/120/150 and 180 min).
  Fructose malabsorption will be determined by creating a hydrogen breath curve for each test day.

SECONDARY OUTCOMES:
Gastrointestinal symptoms | Adjusted GSRS (for a 60 min period) will be used to obtain self-reported gastrointestinal distress at -65 min (before exercise), 0 min (directly after exercise), and at 60/120 and 180 min.
  Gastrointestinal distress (measured through multiple adjusted gastrointestinal symptom rating scale (GSRS) questionnaires).

CONTACTS AND LOCATIONS:
Locations (1):
- Health Futures Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided